CLINICAL TRIAL: NCT05021172
Title: Incorporating ePrognosis to Encourage "Smarter Screening" for Breast and Colorectal Cancer in Older Adults
Brief Title: Incorporating ePrognosis for the Encouragement of Smarter Screening for Breast and Colorectal Cancer in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21051; NCI-2021-08493 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Passport to Health booklet, ePrognosis) (Experimental): Participants receive Passport to Health booklet and complete ePrognosis before scheduled primary care visit.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Participants receive usual care before scheduled primary care visit.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Other: Informational Intervention — Receive Passport to Health booklet
  Arms: Arm I (Passport to Health booklet, ePrognosis)
Other: Questionnaire Administration — Complete ePrognosis
  Arms: Arm I (Passport to Health booklet, ePrognosis)
Other: Survey Administration — Ancillary studies
  Arms: Arm II (usual care)

SUMMARY:
This clinical trial assesses the feasibility and acceptability of a smarter screening intervention for breast and colorectal cancer in older adults. This study aims to learn more about how to support patients and physicians in making cancer screening decisions for older adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Complete development of and refine "Smarter Screening", a multi-component, patient-centered intervention centered around ePrognosis: Cancer Screening to facilitate shared decision-making screening discussions for breast and colorectal cancer in older adults.

II. Assess feasibility and acceptability of the "Smarter Screening" intervention and assess its impact versus usual care on shared decision-making about whether or not to continue breast and colorectal cancer (CRC) screening among multi-ethnic and socioeconomically diverse primary care patients.

EXPLORATORY OBJECTIVES:

I. Impact on breast and CRC screening versus usual care.

II. Risk perception, worry, and a patient-reported measure of decision quality.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive Passport to Health booklet and complete ePrognosis before scheduled primary care visit.

ARM II: Participants receive usual care before scheduled primary care visit.

After completion of study, participants are followed up at 1 week post primary care visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and above
* Ability to understand study procedures and to comply with them for the entire length of the study
* Ability of individual to understand a written informed consent document, and the willingness to sign it
* Have no prior history of cancer
* Scheduled for an upcoming appointment in University of California, San Francisco (UCSF) General Internal Medicine or Women's Health Primary Care clinics
* English-speaking

Exclusion Criteria:

* Contraindication to any study-related procedure or assessment
* Non-English speaking
* Are under the current medical care of either the study primary investigator (PI) or co-investigator (Co-I)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants enrolled | 6 months
  Ability to successfully recruit the target of approximately 40 patients will be determined by the overall number of participants who were screened for enrollment compared to the overall number of participants who were randomized to one of the groups.
Proportion of primary care physicians (PCPs) enrolled | 6 months
  Ability to successfully recruit PCPs will be determined by the overall number of physicians who were contacted compared to the overall number of physicians who actively participated over the course of the study.
Percentage of participants enrolled at 6 months | 6 months
  The investigators aim to attain at least 75% of recruited patients in each arm at the 6 month follow-up.
Proportion of participants who received an ePrognosis report | 6 months
  The proportion of participants who received an ePrognosis report will be reported
Proportion of physicians who utilized the ePrognosis clinician report | 6 months
  All enrolled intervention PCPs will receive a web-based survey after each patient visit to record whether the physicians used and/or discussed ePrognosis in that visit. The proportion of physicians who use the ePrognosis clinician report in their cancer screening counseling with participants/patients will be reported
Responses to Qualitative Acceptability survey | 6 months
  A survey will be provided to PCPs and used to measure acceptability of the ePrognosis report by asking patients and providers to provide feedback about the intervention, including likes and dislikes, and future recommendation of using the report provided.

OTHER OUTCOMES:
Proportion of patients screened for breast cancer | 6 months
  The impact on breast cancer screening versus usual care will be measured by comparing the proportion or participants who were screened for cancers by treatment arm.
Proportion of patients screened for colorectal cancer | 6 months
  The impact on colorectal cancer screening versus usual care will be measured by comparing the proportion or participants who were screened for cancers by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Walsh-Cassidy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No